CLINICAL TRIAL: NCT07128160
Title: The Relationship Between Neuropsychiatric, Radiological Findings and Cortical Inhibition in Patients With Multiple Sclerosis: A Hospital-based Study
Brief Title: Cortical Inhibition in Patients With Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abanoub bassem fikry ramzy, Resident Physician, Department of Neurology and Psychiatry, Assiut University, Assiut University
Other Study IDs: cortical intibition in ms
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple sclerosis: patients with multiple sclerosis
  Interventions: Other: Clinical and Demographic Assessment; Other: Corticospinal Inhibition Assessment; Other: Radiological Assessment

INTERVENTIONS:
Other: Clinical and Demographic Assessment — 1. Expanded Disability Status Scale (EDSS) (Kurtzke, 1983): This scale will be used for neurological disability assessment
  2. Multiple Sclerosis Functional Composite (MSFC): This composite will be used for the assessment of functional performance in patients with MS. It includes: a) Timed 25-foot walk (T25FW), b) Nine-hole peg test (9HPT) for both hands, and c) Paced auditory serial addition test (PASAT).
  3. Toronto Alexithymia Scale (TAS-20): This scale reports Alexithymia. It is a 20-item self-report questionnaire measuring three domains: Difficulty identifying feelings (DIF), Difficulty describing feelings (DDF), and externally oriented thinking (EOT). A score ≥ 61 indicates alexithymia (Bagby, Parker & Taylor, 1994).
  4. Montreal Cognitive Assessment (MoCA), (Nasreddine ZS et al, 2005): a 30-point tool that investigates visuospatial abilities, language, attention, memory, abstraction, and orientation, with scores <26 suggestive of mild cognitive impairment
Other: Corticospinal Inhibition Assessment — Corticospinal inhibition will be evaluated using Transcranial Magnetic Stimulation (TMS) (Ayache et al., 2022; Chalah et al., 2018). All TMS assessments will be conducted according to international safety guidelines. The following parameters will be measured:
  1. Motor Evoked Potentials (MEPs) will be recorded from the abductor pollicis brevis muscle.
  2. Cortical silent period (CSP) will be assessed to measure corticospinal excitability and inhibition.
  3. The interhemispheric inhibition (IHI) is a parameter reflecting the transcallosal GABA-mediated inhibitory activity. It will be obtained at complete muscle rest using figure-of-eight coils (MC-B70; MagVenture), connected with a MagPro_R20 (Medtronic Inc., USA) generator connected to a butterfly coil.
Other: Radiological Assessment — All patients will undergo brain and spinal cord Magnetic Resonance Imaging (MRI) using a 1.5T scanner. Brain MRI sequences include: T1-weighted, T2-weighted, FLAIR, and post-contrast sequences. Spinal MRI (cervical and thoracic) includes T2-weighted and STIR sequences. Radiological assessment focused on:
  * Number and location of T2/FLAIR lesions
  * Presence of contrast-enhancing lesions
  * Degree of brain atrophy (qualitatively)
  * Spinal cord lesion load A neuroradiologist will review MRI findings, blinded to the clinical and neuropsychological data

SUMMARY:
1. To investigate the relationship between corticospinal inhibition and clinical, psychological, and cognitive features in MS patients.
2. To examine the association between corticospinal inhibition and radiological findings, including MRI lesions and white matter damage

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic immune-mediated disorder of the central nervous system (CNS), characterized by demyelinating white matter lesions and diffuse neurodegeneration. These pathological changes lead to variable and unpredictable clinical presentations and disease progression. Beyond motor and sensory deficits, MS is frequently associated with cognitive and emotional disturbances. Cognitive impairment affects 40-70% of patients, particularly in domains such as attention, processing speed, executive functions, and working memory-significantly impacting daily life and quality of care.

Alexithymia, a condition involving difficulty in identifying and describing emotions, externally oriented thinking, and limited imaginative ability, has been reported in a substantial proportion of patients, especially in progressive forms of the disease. It is frequently associated with sleep disturbances, anxiety, and depression.

Fatigue is one of the most burdensome and common symptoms in MS. It may present at any stage and is defined as a persistent lack of physical or mental energy that interferes with daily function. Fatigue may be classified as primary-linked directly to MS pathophysiology-or secondary, due to comorbid conditions, medication effects, or inactivity. Unlike general fatigue, MS-related fatigue is not relieved by rest and has a distinctly disabling nature.

Depression is another prevalent comorbidity, with lifetime prevalence in MS ranging widely. Its development reflects both the psychological burden of chronic disease and neurobiological mechanisms, such as inflammation and demyelination affecting mood circuits.

Given this wide spectrum of motor, cognitive, and emotional manifestations, comprehensive and multidimensional tools are essential for assessing the functional impact of MS. The Multiple Sclerosis Functional Composite (MSFC) is one such standardized, performance-based assessment. It captures core aspects of MS-related disability across three domains: ambulation (Timed 25-Foot Walk, T25FW), upper limb coordination (9-Hole Peg Test, 9HPT), and cognition (Paced Auditory Serial Addition Test, PASAT-3).

Magnetic resonance imaging (MRI) plays a pivotal role in both diagnosis and disease monitoring. Beyond identifying dissemination in time and space, advanced MRI techniques have linked symptom burden-particularly fatigue and cognitive deficits-to microstructural damage in normal-appearing white matter. This suggests that functional disconnection, rather than lesion volume alone, contributes to clinical manifestations.

Transcranial magnetic stimulation (TMS) provides a non-invasive, neurophysiological method to assess corticospinal excitability. When applied to the primary motor cortex, TMS elicits motor-evoked potentials (MEPs) that reflect both direct and trans-synaptic activation of motor pathways, offering insights into cortical inhibition and conduction properties in MS.

Despite advances in neuroimaging and functional assessments, the relationship between corticospinal inhibition and the heterogeneous symptomatology of multiple sclerosis-including fatigue, cognitive dysfunction, and emotional dysregulation-remains underexplored. Few studies have integrated transcranial magnetic stimulation (TMS) with clinical, cognitive, and radiological metrics in a multidimensional framework. This gap limits understanding of the neurophysiological substrates underlying these complex and disabling symptoms.

The present study aims to investigate the relationship between corticospinal inhibition, as assessed by TMS, and the clinical, psychological, cognitive, and radiological profiles of patients with multiple sclerosis. The hypothesis is that altered corticospinal inhibition will correlate with increased fatigue, cognitive dysfunction, alexithymia, and specific MRI abnormalities, reflecting the integrated neurophysiological basis of multiple sclerosis-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of RRMS based on the 2017 McDonald Criteria.
3. Expanded Disability Status Scale (EDSS) score ≤ 6.5.
4. On a stable dose of disease-modifying therapy (DMT) for at least 3 months or naeive patients not use DMT before
5. Free of relapses or steroids treatment (at least 3 months after a relapse or corticosteroid therapy)
6. Ability to give informed consent and complete neuropsychological assessments.

Exclusion Criteria:

1. Presence of other neurological or psychiatric disorders (e.g., major depression, bipolar disorder, schizophrenia).
2. History of alcohol or substance abuse.
3. Contraindications to MRI (e.g., pacemakers, metallic implants) and TMS (i.e., history of seizures, presence of ferromagnetic implants in the head area).
4. Medications known to alter the corticospinal excitability.
5. Severe visual deficit, motor weakness, or intellectual impairment (as per the Mini-Mental State Exam score < 24).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the sample size calculation was performed using EpI-Info 2002 software statistical package designed by World Health Organization (WHO) and by Centers for Disease Control and Prevention (CDC). The sample size was calculated based on the following considerations: 95% confidence level and according to a previous study (Chaves, A. R.,2024). Therefore, resulting sample size of 82 thus sample size increased to 90
  Chaves, A. R., Tremblay, S., Pilutti, L., & Ploughman, M. (2024). Lowered ratio of corticospinal excitation to inhibition predicts greater disability, poorer motor and cognitive function in multiple sclerosis. Heliyon, 10(15).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potential (MEP) | baseline
  Obtained using single-pulse transcranial magnetic stimulation over the primary motor cortex. Latency is defined as the time interval from the TMS pulse to the onset of the muscle response. Longer latencies may indicate impaired corticospinal conduction.
Cortical Silent Period (CSP) | baseline
  Recorded during sustained voluntary muscle contraction using TMS. The silent period is the time during which voluntary electromyographic activity is suppressed following the motor evoked potential. CSP reflects intracortical inhibitory mechanisms.
Interhemispheric Inhibition (IHI) | baseline
  The interhemispheric inhibition (IHI) is a parameter reflecting the transcallosal GABA-mediated inhibitory activity. It will be obtained at complete muscle rest using figure-of-eight coils (MC-B70; MagVenture)

SECONDARY OUTCOMES:
Toronto Alexithymia Scale (TAS-20) | baseline
  A 20-item self-report measure that evaluates difficulty in identifying feelings, difficulty in describing feelings, and externally oriented thinking. Each item is rated on a 5-point Likert scale, with higher scores indicating greater alexithymia.
Fatigue Severity Scale (FSS) | baseline
  A self-reported questionnaire consisting of nine items that assess the impact of fatigue on daily functioning. Each item is scored on a 7-point Likert scale, with higher scores indicating greater fatigue severity.